CLINICAL TRIAL: NCT05241340
Title: A Phase II Clinical Trial of Neoadjuvant Sasanlimab and Stereotactic Body Radiation Therapy as an in Situ Vaccine for Cisplatin-ineligible Muscle Invasive Bladder Cancer
Brief Title: Neoadjuvant Sasanlimab With Radiation as an in Situ Vaccine for Cisplatin-ineligible Muscle Invasive Bladder Cancer
Acronym: RAD-VACCINE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Raj Satkunasivam, Associate Professor, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00032433
Record Dates: First submitted 2022-01-19; First posted 2022-02-15 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Urothelial Carcinoma Bladder
Keywords: Bladder Cancer; Muscle Invasive Bladder Cancer; Immune Checkpoint Inhibitor; Immunotherapy; Urothelial Carcinoma of the Bladder; Urologic neoplasms; Neoadjuvant therapy; Radiation; Stereotactic Body Radiation Therapy; Urinary Bladder Diseases; Urologic Diseases; Sasanlimab; Antineoplastic agents; Antineoplastic agents, Immunological
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urologic Neoplasms; Urinary Bladder Diseases; Urologic Diseases | interventions — Immune Checkpoint Inhibitors; Radiosurgery; Cystectomy; Urinary Diversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open arm (Experimental): All patients will receive study interventions (sasanlimab and SBRT) and standard-of-care radical cystectomy.
  Interventions: Drug: Sasanlimab; Radiation: Stereotactic Body Radiation Therapy; Procedure: Radical Cystectomy + pelvic lymph node dissection + urinary diversion

INTERVENTIONS:
Drug: Sasanlimab — Sasanlimab (PF-06801591) is a recombinant humanized monoclonal antibody (immunoglobulin gamma-4 with kappa light chains, IgG4 kappa) directed against programmed death 1 (PD-1). Manufactured by Pfizer, Inc.
  Other Names: PF-06801591; PD-1 Inhibitor
Radiation: Stereotactic Body Radiation Therapy — This current study is designed to deliver a biologically equivalent dose of 43.2Gy using a strategy of HD hypo-fractionated radiation therapy 8Gy x 3 in combination with Sasanlimab
Procedure: Radical Cystectomy + pelvic lymph node dissection + urinary diversion — This will include a cysto-prostatectomy in males or a radical cystectomy with anterior exenteration in females, bilateral pelvic lymph node dissection, and creation of a urinary diversion (ileal conduit, Indiana pouch or orthotopic neo-bladder). Robotic assisted or open surgery will be permitted.
  Because there is currently equipoise regarding standard or extended template pelvic lymph node dissection, the limits of node dissection will not be protocol mandated. In the standard template, nodal packets will include the common iliac, external iliac, internal iliac (or hypogastric) and obturator nodes. Patients receiving an extended template will have the standard nodes with the addition of the para-aortic, para-caval, pre-sacral, and pre-sciatic node packets. The decision for urinary diversion is multifactorial involving patient factors (e.g., adequate renal function) and preference; thus, it will be made on a case-by-case basis.

SUMMARY:
This is a prospective, single-institution, single-arm, phase II clinical trial that tests a novel strategy of neoadjuvant Sasanlimab, an immune checkpoint inhibitor (ICI), in combination with stereotactic body radiation therapy as an in-situ vaccination in patients, who are ineligible to receive cisplatin-based chemotherapy and undergoing radical cystectomy for muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
Patients with cT2-T4a, N0, M0 urothelial bladder carcinoma (UBC) after transurethral resection of the bladder will receive 2 doses of sasanlimab (PF-06801591) at the dose of 300mg subcutaneously, followed by 3 doses of radiation (8Gy x 3) prior to surgery (radical cystectomy). Cystectomy will be planned to be done within 6 weeks of the last dose of sasanlimab.

Pathologic complete response (pT0) is the primary endpoint, in addition to a safety lead-in endpoint consisting of a composite outcome of feasibility and safety.

Exploratory biomarker analysis on tissue/blood samples will include genomic and immune-system profiling in tumor and blood before and after sasanlimab/radiation therapy, and after radical cystectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent
2. Age ≥ 18 years
3. ECOG Eastern Cooperative Oncology Group performance status 0-2
4. Predominant (>50%) urothelial carcinoma histology
5. Muscle-invasive bladder cancer (cT2-4a, cN0, cM0)
6. Decline/refuse OR Ineligible to receive cisplatin-based Neoadjuvant Chemotherapy due to at least one of the following criteria:

   a. Creatinine clearance less than 60 mL/min b. Eastern Cooperative Oncology Group performance status of ≥ 2 c. Grade ≥ 2 hearing loss d. Grade ≥ 2 neuropathy
7. Adequate Bone Marrow Function (without hematopoietic growth factor support within 14 days prior to study screening), defined as:

   a. Absolute neutrophil count (ANC) ≥1,500/mm3 or ≥1.5 x 109/L b. Platelets ≥100,000/mm3 or 100 x 109/L c. Hemoglobin ≥9 g/dL (≥5.6 mmol/L)
8. Adequate renal function defined by an estimated creatinine clearance ≥30 mL/min according to the Cockcroft Gault formula or by 24-hour urine collection for creatinine clearance.
9. Adequate liver function, including:

   a. Aspartate and alanine aminotransferase (AST and ALT) ≤ 2.5 × the upper normal limit range (ULN) b. Total serum bilirubin ≤ 1.5 x ULN
10. Able to give informed consent and patient is willing and able to comply with scheduled study visits and treatment plan
11. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other procedures.
12. Meeting the following criteria for sex specific considerations:

<!-- -->

1. Males - for the duration of study and for at least 6 months after the last dose of study drug (Sasanlimab):

   1. Refrain from donating sperm and be abstinent from intercourse OR Agree to use male condom and also consider the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant
2. Females:

   a) Eligible to participate if not pregnant or breast feeding AND Is not a woman of childbearing potential (WOCBP) OR Is a WOCBP and is using a contraceptive method that is highly effective (failure rate of < 1% per year), with low user dependency during the during the study treatment and for at least 6 months after the last dose of study drug (Sasanlimab) b) A WOCBP must have a negative, highly sensitive (at least 25 IU/mL) pregnancy test by urine or serum testing within 24 hours before the first dose of study drug (Sasanlimab). In cases where the urine test cannot be confirmed to be negative, a serum pregnancy test will be used.

Exclusion Criteria:

1. Lymphadenopathy (>1cm short-axis measurement on CT/MRI Imaging or biopsy proven)
2. Metastatic disease
3. Prior systemic chemotherapy for bladder cancer (however, may have had intra-vesical chemotherapy such as gemcitabine, docetaxel or mitomycin-C)
4. Prior treatment with systemic anti-cancer investigational agent
5. Other malignancy within 2 years prior to study screening, or active malignancy except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix, or low-grade (Gleason 6 or below) prostate cancer on surveillance without any plans for treatment intervention (e.g., surgery, radiation, or castration) or other concurrent malignancy felt by the investigator has a very low likelihood to become metastatic
6. Previous radiation therapy to the bladder
7. Active or history of autoimmune disease which may deteriorate when receiving immune checkpoint blockade.

   1. These autoimmune conditions include but are not limited to limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis
   2. Participants with diabetes type I, vitiligo, psoriasis, or hypo or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
8. Severe active infections (e.g., pulmonary tuberculosis) requiring systemic therapeutic oral or IV antibiotics within 2 weeks prior to study entry.
9. Clinically significant, multiple or severe drug allergies, intolerance to topical corticosteroids
10. Current unstable liver or biliary disease, defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.

    * NOTE: Stable chronic liver disease (including Gilbert's syndrome, asymptomatic gallstones, and chronic stable hepatitis B or C -e.g., presence of hepatitis B surface antigen [HBsAg] or positive hepatitis C antibody test result at screening) is acceptable.
11. Active, uncontrolled HIV/AIDS infection (well-controlled HIV patients may be allowed).
12. Prior immunotherapy with anti PD-1, anti PD-L1, anti PD-L2, or anti cytotoxic T- lymphocyte-associated antigen-4 (CTLA-4) antibody. Note: prior intra-vesical BCG therapy is acceptable.
13. Prior treatment with immune-stimulatory agents including interleukin (IL)-2, IL-15, interferon (INF)- γ.
14. Vaccination within 4 weeks from study screening and while on study treatment unless administration of inactivated vaccines.
15. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
16. Clinically significant (active) cardiovascular disease including the following: cerebral vascular accident/stroke <6 months prior to screening; myocardial infarction <6 months prior to screening; unstable angina; congestive heart failure (≥New York Heart Association Classification Class III); or serious cardiac arrhythmia (uncontrolled, clinically significant) requiring medication.
17. Q-T interval corrected for heart rate (QTc) >450 msec for male participants or QTc >470 msec for female participants or QTc >480 msec in participants with right bundle branch block
18. Prior organ transplantation or allogenic stem cell transplantation.
19. Known history of: immune-mediated colitis, inflammatory bowel disease, pneumonitis, or pulmonary fibrosis.
20. Patients with intolerance to or who have had a severe (Grade ≥3) allergic or anaphylactic reaction to antibodies or infused therapeutic proteins
21. Pregnant female patients; breastfeeding female patients; male patients able to father children and female patients of childbearing potential who are unwilling or unable to use a highly effective method(s) of contraception as outlined in this protocol for at least 6 months after the last dose of Sasanlimab (PF-06801591)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome for Feasibility and Safety | From date of registration to date of death due to any cause, assessed up to 4 weeks after radical cystectomy
  Combination of Sasanlimab and SBRT will be deemed both feasible and safe (composite outcome) if, after the treatment of 10 patients, ≥ 7 of 10 patients meet all of the following feasibility criteria:
  1. Receive at least 1 dose of 2 of Sasanlimab
  2. Receive at least 2 of 3 fractions SBRT
  3. Undergo radical cystectomy RC within 4 weeks of completing therapy (after end of cycle 2)
  and meet all of the safety criteria, defined as not experiencing any following Common Terminology Criteria for Adverse Events (CTCAE) toxicities up to 4 weeks after the completion of radical cystectomy:
  1. Hematologic toxicity ≥ Grade 4
  2. Non-hematologic toxicity ≥ Grade 3
  3. Non-hematologic toxicity ≥ Grade 2 lasting >1 week (except alopecia, emesis, and laboratory abnormalities)
Clinical benefit rate defined as pathologic complete response (pT0) | At time of radical cystectomy
  Proportion of patients experiencing pathologic complete response (pT0) after the study treatment followed by radical cystectomy.

SECONDARY OUTCOMES:
Incidence of adverse events graded by NCI CTCAE version 5.0 | From date of registration to date of death due to any cause, assessed up to 12 weeks after radical cystectomy
  Graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Incidence of major surgical complications graded by Clavien-Dindo Scale | From date of radical cystectomy to date of death, assessed up to 30 days following surgery
  Clavien-Dindo scale is widely utilized for grading adverse events (i.e. complications) that may occur as a result of surgical procedures.
  The severity of the complication increases from grade 1 to grade 5.
Health Related Quality of Life for Patients with T2-T4 muscle invasive bladder cancer | From date of registration to date of death due to any cause, assessed up to 24 months after radical cystectomy
  Patient's health related quality of life survey on 30 items including urinary symptoms, sexual function, urostomy issues, catheter use, and body image will be assessed by The European Organization for Research and Treatment of Cancer (EORTC) QOL C30-BLM 30, in order to assess changes in patient-reported quality of life at baseline and changes.
  Each item is scored on a 4 point scale, with a higher score reflecting a better quality of life.
Overall survival (OS) | From date of registration to date of death due to any cause, assessed up to 24 months after radical cystectomy
  Overall Survival is defined as the duration of time from the date of treatment initiation that a patient is still alive.
Recurrence free survival (RFS) | From date of registration to date of death due to any cause, assessed up to 24 months after radical cystectomy
  RFS is defined as the time from surgery and study treatment to recurrence or death, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Raj Satkunasivam, MD, Principal Investigator — Houston Methodist Hospital, Houston Methodist Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Satkunasivam R, Lim K, Teh BS, Guzman J, Zhang J, Farach A, Chen SH, Wallis CJ, Efstathiou E, Esnaola NF, Sonpavde GP. A phase II clinical trial of neoadjuvant sasanlimab and stereotactic body radiation therapy as an in situ vaccine for cisplatin-ineligible MIBC: the RAD VACCINE MIBC trial. Future Oncol. 2022 Aug;18(25):2771-2781. doi: 10.2217/fon-2022-0380. Epub 2022 Jun 15. PMID 35703113